CLINICAL TRIAL: NCT00945945
Title: A Phase 3b Study to Assess the Efficacy of Duloxetine 60 mg Once Daily Compared With Placebo on the Reduction of Pain Caused by Osteoarthritis of the Knee, in a 13-week, Double-blind, Randomized Study
Brief Title: A Study of Duloxetine in Patients With Osteoarthritis Knee Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13214; F1J-MC-HMGP (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Results first posted 2011-03-08 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-02

CONDITIONS: Osteoarthritis Knee Pain
Keywords: Osteoarthritis, Knee; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DLX30-PLA (Experimental): Per the protocol, patients randomized to the duloxetine group were to receive duloxetine for the entire 13-week acute treatment period. Patients were to start at a 30 mg daily (QD) dose of duloxetine for 1 week, then increase to 60 mg QD of duloxetine for the following 12 weeks. However, due to a study drug labeling error, patients randomized to this group received 30 mg of duloxetine for the initial 1-week, but received placebo instead of receiving 60 mg QD of duloxetine for the next 12 weeks. The resulting unintended, mixed treatment group was labeled as DLX30-PLA throughout this document. Per protocol, the last week of the study (week 14) was intended to be a 1-week taper period. Patients in this treatment group were to receive 30 mg QD of duloxetine during that week, and that did occur per protocol.
  Interventions: Drug: Duloxetine (DLX); Drug: Placebo (PLA)
- PLA-DLX60 (Placebo Comparator): Per the protocol, patients randomized to the placebo group were to receive placebo for the entire 13-week acute treatment period. Patients were to start on placebo for the first week, then continue on placebo for the following 12 weeks. However, due to a study drug labeling error, patients in this group received placebo for the initial 1-week, but received 60 mg QD of duloxetine instead of receiving placebo for the next 12 weeks. The resulting unintended, mixed treatment group was labeled as PLA-DLX60 throughout this document. Per protocol, the last week of the study (week 14) was intended to be a 1-week taper period. Patients in this treatment group were to receive placebo that week, and that did occur per protocol.
  Interventions: Drug: Duloxetine (DLX); Drug: Placebo (PLA)

INTERVENTIONS:
Drug: Duloxetine (DLX) — dose daily by mouth
  Other Names: LY248686; Cymbalta
Drug: Placebo (PLA) — Placebo Comparator daily by mouth

SUMMARY:
The primary purpose of this study is to determine if duloxetine 60 mg once daily (QD) reduces pain severity in patients with osteoarthritis (OA) knee pain compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients with osteoarthritis knee pain for greater than or equal to 14 days of each month for 3 months prior to study entry.
* Have a rating of greater than or equal to 4 on the BPI average pain item (Question 3 of the Brief Pain Inventory [BPI] modified short form) at screening and randomization

Exclusion Criteria:

* Have had any previous exposure to duloxetine.
* Have any previous diagnosis of psychosis, bipolar disorder, or schizoaffective disorder.
* Have Major Depression Disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, as assessed by the Mini International Neuropsychiatric Interview (Sheehan et al. 1998), or diagnosed within the past year.
* Have a history of substance abuse or dependence within the past year, excluding nicotine and caffeine.
* Are taking any excluded medications that cannot be discontinued at screening visit.
* Have current or pending disability compensation or litigation issues that may compromise response to treatment, in the opinion of the investigator.
* Have had treatment with a monoamine oxidase inhibitor (MAOI) within 14 days of randomization or the potential need to use an MAOI during the study or within 5 days of discontinuation of study drug.
* Have a positive urine drug screen for any substance of abuse or excluded medication.
* Are pregnant or breast-feeding.
* Have serious cardiovascular, hepatic, renal, respiratory, or hematologic illness, or other medical or psychiatric condition that, in the opinion of the investigator, would compromise participation or be likely to lead to hospitalization during the course of the study.
* Have a history of recurrent seizures other than febrile seizures.
* Are judged by the investigator to be at suicidal risk.
* Have uncontrolled narrow-angle glaucoma.
* Have acute liver injury (such as hepatitis) or severe cirrhosis (Child- Pugh Class C).
* Have known hypersensitivity to duloxetine or any of the inactive ingredients or patients with frequent or severe allergic reactions to multiple medications.
* Have frequent falls that could result in hospitalization or could compromise response to treatment.
* Have a confounding painful condition that may interfere with assessment of the index joint, that is, knee. (Knee pain should be the predominant pain. Mild OA pain of other joints is allowed.)
* Have a diagnosis of inflammatory arthritis (that is, rheumatoid arthritis) or an autoimmune disorder (excluding inactive Hashimoto's thyroiditis).
* Have received intraarticular hyaluronate or steroids, joint lavage, or other invasive therapies to the knee in the past 3 months.
* Have had knee arthroscopy of the index knee within the past year or joint replacement of the index knee at anytime.
* Have surgery planned during the study for the index joint.
* Have a body mass index (BMI) over 40.
* Use of acupuncture, chiropractic maneuvers, transcutaneous electrical nerve stimulation (TENS), or similar procedures aimed to relieve any kind of pain.
* Patients who are anticipated by the investigator to require use of analgesic agents including but not limited to non-steroidal anti-inflammatory drugs(NSAIDs), acetaminophen/paracetamol, and opioids, or other excluded medication for the duration of the study.
* Are unwilling or unable to comply with the data collection method used to record their patient rated outcome data.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (26):
- United States (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Montgomery, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Spring Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Morton Grove, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Prairie Village, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Toledo, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Myrtle Beach, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Lake Jackson, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Clinton, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Oregon, Wisconsin
- Germany (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Rhaunen
- Greece (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Heraklion
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Kifissia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Marousi Attikis
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Thessaloniki
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Ponce, Puerto Rico
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Bucharest, Romania
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Moscow, Russia
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, A Coruña
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Getafe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Madrid
- Sweden (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Malmo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Uddevalla

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to a study drug labeling error which led to a treatment crossover, the intended comparisons for group-level differences between duloxetine and placebo cannot be made. The results from comparisons of mixed-treatment groups are presented for primary efficacy and safety outcomes.
Period: Overall Study
Arm/Group | DLX30-PLA | PLA-DLX60
Started | 207 | 217
Completed | 171 | 162
Not Completed | 36 | 55
Not completed — Adverse Event | 15 | 35
Not completed — Withdrawal by Subject | 7 | 10
Not completed — Lost to Follow-up | 4 | 5
Not completed — Lack of Efficacy | 6 | 2
Not completed — Protocol Violation | 4 | 2
Not completed — Entry Criteria Not Met | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DLX30-PLA | PLA-DLX60 | Total
Number analyzed (Participants) | 207 | 217 | 424
Age Continuous [Mean (Standard Deviation); unit: years] | 63.40 (9.90) | 64.18 (10.06) | 63.80 (9.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 141 | 288
  Male | 60 | 76 | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 27 | 53
  Not Hispanic or Latino | 181 | 190 | 371
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 13 | 21
  White | 196 | 203 | 399
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 81 | 92 | 173
  Puerto Rico | 3 | 4 | 7
  Greece | 13 | 11 | 24
  Spain | 25 | 23 | 48
  Romania | 16 | 19 | 35
  Russian Federation | 33 | 32 | 65
  Germany | 18 | 19 | 37
  Sweden | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 13 Week Endpoint (Baseline Observation Carried Forward [BOCF]) in Brief Pain Inventory (BPI) "24-Hour Average Pain" Item (Question 3) of the BPI-Modified Short Form Score
Description: A self-reported measure of the severity of pain based on the average pain over 24-hours. Severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). BOCF endpoint was defined as the baseline value for participants discontinued during acute phase, and defined as the last non-missing observation in the treatment phase for all other randomized participants. Due to the nature of a study drug labeling error which led to a treatment crossover (see Arms), data from protocol-defined treatment groups were compromised. The results from each mixed-treatment group are presented.
Time Frame: Baseline, 13 weeks
Population: Number of randomized participants with a non-missing baseline and BOCF endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DLX30-PLA | PLA-DLX60
Number analyzed (Participants) | 207 | 217
units on a scale
  Baseline | 6.00 (1.28) | 6.10 (1.31)
  Change from Baseline to Endpoint (BOCF) | -1.93 (2.23) | -2.34 (2.30)
Statistical Analysis 1: Comparison: DLX30-PLA vs PLA-DLX60; Test type: Superiority or Other; p = 0.105, ANCOVA — P-value for Change from Baseline to Endpoint (BOCF); Main Effect Model: Change = Treatment + Pooled Investigator + Baseline (Type III sums of squares); Least Squares Mean Difference = 0.34, 95% CI 2-sided [-0.07 to 0.75] — Least Squares Mean Difference = DLX30-PLA minus PLA-DLX60

2. Secondary Outcome: Number of Participants With Suicidal Behaviors and Ideations From the Columbia Suicide Severity Rating Scale
Description: C-SSRS: scale capturing occurrence, severity, and frequency of suicide-related thoughts and behaviors. Number of patients with suicidal behaviors and ideations are provided. Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation: a "yes" answer to any one of 5 suicidal ideation questions, which includes wish to be dead, and 4 different categories of active suicidal ideation.
Time Frame: Baseline through 13 weeks
Population: All randomized participants.
Measure: Number; unit: participants
Arm/Group | DLX30-PLA | PLA-DLX60
Number analyzed (Participants) | 207 | 217
participants
  Ideation: Wish to be dead | 1 | 0
  Ideation: Non-specific active suicidal thoughts | 0 | 0
  Ideation: Active suicidal ideation without intent | 0 | 0
  Ideation: Active suicidal ideation with intent | 0 | 0
  Ideation:Active suicidal ideation with plan to act | 0 | 0
  Behavior: Preparatory acts or behavior | 0 | 0
  Behavior: Aborted attempt | 0 | 0
  Behavior: Interrupted attempt | 0 | 0
  Acts: Non-fatal suicide attempt | 0 | 0
  Acts: Completed suicide | 0 | 0

3. Secondary Outcome: Mean Change From Baseline to Endpoint (13 Week) in Patient's Global Impressions of Improvement Score
Description: A scale that measures the patient's perception of improvement at the time of assessment compared with the start of treatment. The score ranges from 1 (very much better) to 7 (very much worse). Due to the nature of a study drug labeling error and the resultant treatment crossover (see Arms), the data from both protocol-defined treatment groups were compromised, and the intended comparisons for differences between those treatment groups are considered unevaluable. Secondary efficacy results from the 2 mixed-treatment groups are not presented.
Time Frame: Baseline, 13 weeks
Measure: Mean (Standard Deviation); unit: participants
Arm/Group | DLX30-PLA | PLA-DLX60
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Mean Change From Baseline to Endpoint (13 Week) in Western Ontario McMaster Universities (WOMAC) Index Score
Description: The WOMAC index (pain, stiffness, physical function subscales) was completed by the patient. The index has 24 questions. Each question is answered using a 5-point Likert scale (0 to 4). The Total score has a range from 0 (none) to 96 (extreme). Due to the nature of a study drug labeling error and the resultant treatment crossover (see Arms), data from both protocol-defined treatment groups were compromised, and the intended comparisons for differences between those treatment groups are considered unevaluable. Secondary efficacy results from the 2 mixed-treatment groups are not presented.
Time Frame: baseline, 13 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DLX30-PLA | PLA-DLX60
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Mean Change of Total Score From Baseline to Endpoint (13 Week) of Brief Pain Inventory-Severity (BPI-S) Scale
Description: Self-reported scale measuring pain severity. Severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). Four questions assess worst pain, least pain, and average pain in the past 24 hours, and pain right now. Total score ranges from 0-40. Due to the nature of a study drug labeling error and resultant treatment crossover, data from both protocol-defined treatment groups were compromised, and the intended comparisons for differences between those treatment groups are considered unevaluable. Secondary efficacy results from the 2 mixed-treatment groups are not presented.
Time Frame: Baseline, 13 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DLX30-PLA | PLA-DLX60
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Mean Change of Total Score From Baseline to Endpoint (13 Week) in Brief Pain Inventory- Interference Score
Description: Interference scores range from 0 (does not interfere) to 10 (completely interferes) on 7 questions assessing interference of pain for general activity, mood, walking ability, normal work, relations with others, sleep, and enjoyment of life. Total score ranges from 0-70. Due to the nature of study drug labeling error and resultant treatment crossover, data from both protocol-defined treatment groups were compromised, and intended comparisons for differences between those treatment groups are considered unevaluable. Secondary efficacy results from the 2 mixed-treatment groups are not presented.
Time Frame: Baseline, 13 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DLX30-PLA | PLA-DLX60
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Mean Change of Total Score From Baseline to Endpoint (13 Week) in Clinical Global Impressions of Severity (CGI-S)
Description: Measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). Due to the nature of a study drug labeling error and the resultant treatment crossover (see Arms), the data from both protocol-defined treatment groups were compromised, and the intended comparisons for differences between those treatment groups are considered unevaluable. Secondary efficacy results from the 2 mixed-treatment groups are not presented.
Time Frame: Baseline, 13 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DLX30-PLA | PLA-DLX60
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Mean Change of Total Score From Baseline to Endpoint(13 Week) in Intermittent and Constant Osteoarthritis Pain: Knee Version
Description: An 11-item questionnaire to individually and jointly assess intermittent and constant pain. Questions assess intensity and impact of pain on activity and emotion. Each item is scored from 0 to 4; higher values indicate higher severity. Total Pain score ranges from 0-44. Due to the nature of study drug labeling error and resultant treatment crossover, data from both protocol-defined treatment groups were compromised, and intended comparisons for differences between those treatment groups are considered unevaluable. Secondary efficacy results from the 2 mixed-treatment groups are not presented.
Time Frame: Baseline, 13 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DLX30-PLA | PLA-DLX60
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Mean Change of Total Score From Baseline to Endpoint (13 Week) in Profile of Mood States- Brief Form (BPOMS)
Description: BPOMS measures mood states and has 6 factors: tension-anxiety, depression-dejection, anxiety-hostility, fatigue, confusion, and vigor. Item scores: 0 (not at all) to 4 (extremely). Each factor scores range from 0-20. Total score = sum of all factor scores minus vigor score. Due to nature of study drug labeling error and resultant treatment crossover, data from both protocol-defined treatment groups were compromised, and intended comparisons for differences between those treatment groups are considered unevaluable. Secondary efficacy results from the 2 mixed-treatment groups are not presented.
Time Frame: Baseline, 13 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DLX30-PLA | PLA-DLX60
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Mean Change of Total Score From Baseline to Endpoint (13 Week) in European Quality of Life Questionnaire (EQ-5D)
Description: Patients rate their health state in 5 domains: mobility, self-care, usual activities, pain, and mood. Score between 1-3 is generated for each domain which is mapped to single index score. Index ranges between 0-1; higher scores indicate better health perceived by patient. Due to nature of study drug labeling error and resultant treatment crossover, data from both protocol-defined treatment groups were compromised, and intended comparisons for differences between those treatment groups are considered unevaluable. Secondary efficacy results from the 2 mixed-treatment groups are not presented.
Time Frame: Baseline, 13 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DLX30-PLA | PLA-DLX60
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Mean Change From Baseline to Endpoint (13 Week) in 36-item Short-Form Health Survey
Description: Self-reported questionnaire with 36 questions covering 8 health domains. Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale, with higher scores indicating better health status or functioning. Due to the nature of a study drug labeling error and the resultant treatment crossover (see Arms), the data from both protocol-defined treatment groups were compromised, and the intended comparisons for differences between those treatment groups are considered unevaluable. Secondary efficacy results from the 2 mixed-treatment groups are not presented.
Time Frame: Baseline, 13 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DLX30-PLA | PLA-DLX60
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | DLX30-PLA | PLA-DLX60
Serious Adverse Events (participants affected / at risk) | 3/207 | 2/217
Other Adverse Events (participants affected / at risk) | 105/207 | 143/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DLX30-PLA (N=207) | PLA-DLX60 (N=217)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Neuroborreliosis (Infections and infestations) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DLX30-PLA (N=207) | PLA-DLX60 (N=217)
Constipation (Gastrointestinal disorders) | 7 (7) | 12 (12)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 14 (14)
Dry mouth (Gastrointestinal disorders) | 11 (11) | 19 (20)
Nausea (Gastrointestinal disorders) | 21 (21) | 41 (43)
Fatigue (General disorders) | 3 (3) | 17 (17)
Nasopharyngitis (Infections and infestations) | 16 (18) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 16 (16)
Dizziness (Nervous system disorders) | 6 (6) | 26 (26)
Headache (Nervous system disorders) | 19 (21) | 21 (23)
Somnolence (Nervous system disorders) | 4 (4) | 11 (11)
Insomnia (Psychiatric disorders) | 4 (4) | 13 (15)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (3) | 13 (13)

LIMITATIONS AND CAVEATS:
Due to a package labeling error, study drug was incorrectly administered to all patients in both treatment groups. This compromised the integrity of the entire study and rendered planned comparisons between duloxetine and placebo invalid.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days